CLINICAL TRIAL: NCT03283319
Title: Randomized, Double-Blinded, Phase 2 Study to Assess Safety and Immunogenicity of Panblok H7 Vaccine at Three Antigen Dose Levels Adjuvanted With AS03® or MF59®
Brief Title: Panblok H7 Vaccine Adjuvanted With AS03 or MF59
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Collaborators: Rho, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BP-I-17-002; HHSO100201400004I (Other Grant/Funding Number: BARDA); TO# HHSO10033001T (Other Grant/Funding Number: BARDA)
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Results first posted 2019-09-25 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Influenza, Human
Keywords: Influenza; human; Influenza in Birds; Orthomyxoviridae Infections; RNA Virus Infections; Virus Diseases; Respiratory Tract Infections; Respiratory Tract Diseases; MF59; AS03; Adjuvants; Immunologic
MeSH Terms: conditions — Influenza, Human; Influenza in Birds; Orthomyxoviridae Infections; RNA Virus Infections; Virus Diseases; Respiratory Tract Infections; Respiratory Tract Diseases | interventions — MF59 oil emulsion

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of the six treatment groups at Day 1 and will receive the assigned dose of antigen and adjuvant on Day 1 and Day 29.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 3.75 ug Panblok H7 plus AS03 (Experimental): Participants dosed intramuscularly (IM) on Days 1 and 29 with 3.75 ug Panblok H7 plus AS03
  Interventions: Biological: 3.75 ug Panblok H7; Biological: AS03
- 7.5 ug Panblok H7 plus AS03 (Experimental): Participants dosed intramuscularly (IM) on Days 1 and 29 with 7.5 ug Panblok H7 adjuvanted with AS03
  Interventions: Biological: 7.5 ug Panblok H7; Biological: AS03
- 15 ug Panblok H7 plus AS03 (Experimental): Participants dosed intramuscularly (IM) on Days 1 and 29 with 15 ug Panblok H7 adjuvanted with AS03
  Interventions: Biological: 15 ug Panblok H7; Biological: AS03
- 3.75 ug Panblok H7 plus MF59 (Experimental): Participants dosed intramuscularly (IM) on Days 1 and 29 with 3.75 ug Panblok H7 adjuvanted with MF59
  Interventions: Biological: 3.75 ug Panblok H7; Biological: MF59
- 7.5 ug Panblok H7 plus MF59 (Experimental): Participants dosed intramuscularly (IM) on Days 1 and 29 with 7.5 ug Panblok H7 adjuvanted with MF59
  Interventions: Biological: 7.5 ug Panblok H7; Biological: MF59
- 15 ug Panblok H7 plus MF59 (Experimental): Participants dosed intramuscularly (IM) on Days 1 and 29 with 15 ug Panblok H7 adjuvanted with MF59
  Interventions: Biological: 15 ug Panblok H7; Biological: MF59

INTERVENTIONS:
Biological: 3.75 ug Panblok H7 — 0.5 mL recombinant Panblok H7 influenza vaccine antigen 15 ug/mL.
  Arms: 3.75 ug Panblok H7 plus AS03; 3.75 ug Panblok H7 plus MF59
Biological: 7.5 ug Panblok H7 — Mix 0.5 mL recombinant Panblok H7 influenza vaccine antigen 30 ug/mL.
  Arms: 7.5 ug Panblok H7 plus AS03; 7.5 ug Panblok H7 plus MF59
Biological: 15 ug Panblok H7 — Mix 0.5 mL recombinant Panblok H7 influenza vaccine antigen 60 ug/mL.
  Arms: 15 ug Panblok H7 plus AS03; 15 ug Panblok H7 plus MF59
Biological: MF59 — 0.5 mL MF59 (39 mg squalene/mL ) adjuvant.
  Arms: 15 ug Panblok H7 plus MF59; 3.75 ug Panblok H7 plus MF59; 7.5 ug Panblok H7 plus MF59
Biological: AS03 — 0.5 mL AS03 (42.4 mg squalene/mL ) adjuvant.
  Arms: 15 ug Panblok H7 plus AS03; 3.75 ug Panblok H7 plus AS03; 7.5 ug Panblok H7 plus AS03

SUMMARY:
The main purpose of this study is to assess the safety and ability of a Panblok H7 influenza vaccine adjuvanted with AS03 or MF59 to generate an immune response after 2 doses separated by 28 days. Three different antigen dose levels of Panblok H7 will be tested.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, phase 2 study to assess safety and immunogenicity of Panblok H7 vaccine at three antigen dose levels (3.75, 7.5, and 15 μg) adjuvanted with AS03 or MF59. The main purpose of this study is to assess the safety and ability of the recombinant Panblok H7 influenza vaccine adjuvanted with AS03 or MF59 to generate an immune response after 2 doses separated by 28 days in healthy males and nonpregnant females, aged 18 to 49 years, inclusive. The expected study duration is approximately 13.5 months per participant.

ELIGIBILITY:
Inclusion Criteria:

1. Male or nonpregnant female 18 to 49 years of age, inclusive, at the time of the first study vaccination.
2. Provide written informed consent prior to the initiation of any study-related procedures.
3. Are able to understand and comply with planned study procedures.
4. Have a stable health status based on site investigator's clinical judgment, as established by physical examination, vital signs, and medical history.
5. Have access to a consistent and reliable means of telephone contact, which may be in the home, workplace, or by personal mobile electronic device.
6. Agree to stay in contact with the study site for the duration of the study, have no current plans to move from the study area, and agree to provide updated contact information as necessary.

Exclusion Criteria:

1. Have had a prior severe reaction to any influenza vaccine or have a known allergy to squalene-based adjuvants.
2. Women who are pregnant or breast feeding. Women of childbearing potential must have a negative urine pregnancy test at screening and within 24 hours prior to each vaccination.

   Women of childbearing potential are defined as postmenarcheal and premenopausal females capable of becoming pregnant. This does not include females who meet any of the following conditions: menopausal >12 months, tubal ligation >12 months, bilateral salpingo-oophorectomy, or hysterectomy.
3. Women of childbearing potential who refuse to use an acceptable method of birth control from screening to Day 50 (Visit 7) or, if sexually active with a male partner, who have not used a reliable birth control method during the 2 months prior to screening.

   Adequate contraception is defined as a contraceptive method with a failure rate of less than 1% per year when used consistently and correctly and when applicable, in accordance with the product label, for example: abstinence from penile-vaginal intercourse; oral contraceptives, either combined or progestogen alone; injectable progestogen; implants of etonogestrel or levonorgestrel; estrogenic vaginal ring; percutaneous contraceptive patches; intrauterine device or intrauterine system; male partner sterilization at least 6 months prior to the female participant's Screening Visit, and this male is the sole partner for that participant (the information on the male partner's sterility can come from the site personnel's review of the participant medical records or interview with the participant on her medical history); male condom combined with a vaginal spermicide (foam, gel, film, cream, or suppository); male condom combined with a female diaphragm, either with or without a vaginal spermicide (foam, gel, film, cream, or suppository).
4. Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months, or plans to receive immunosuppressive therapy/cytotoxic treatment during study participation.
5. Have an active neoplastic disease or a history of any hematologic malignancy. However, participants with superficial skin cancer who do not require intervention other than local excision are not excluded.
6. Have long-term use (≥14 consecutive days) of glucocorticoids including oral or parenteral prednisone or prednisone equivalent (>20 mg total dose per day) or high-dose inhaled steroids (>800 µg/day of beclomethasone dipropionate or equivalent) within 1 month prior to screening in this study. However, participants on low-dose inhaled steroids (≤800 µg/day of beclomethasone dipropionate or equivalent) or topical steroids are not excluded.
7. History of schizophrenia, bipolar disease, psychosis, or severe personality disorder.
8. History of hospitalization for psychiatric illness, attempted suicide, or having been deemed a danger to self or others within the past 10 years.
9. Have received immunoglobulin or other blood product (with the exception of Rho[D] immune globulin) within the 3 months prior to screening in this study.
10. Have received any live vaccines within 4 weeks or inactivated or recombinant protein vaccines within 2 weeks prior to screening in this study or plan to receive such vaccines (including seasonal influenza vaccines) from screening through 21 days following the second dose of the study vaccine (Screening Visit through Day 50).
11. Have an acute or chronic medical condition that, in the opinion of the site investigator, would render vaccination unsafe or would interfere with the evaluation of responses. This includes all PIMMCs such as Guillain Barré syndrome, narcolepsy, and current or history of autoimmune or chronic inflammatory disease.
12. Have an acute illness, including body temperature greater than 100.4°F, at screening, immediately prior to each vaccination or, per participant report, within 3 days prior to each vaccination in this study.
13. Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to screening in this study or expect to receive an experimental agent during the study period.
14. Are participating or plan to participate in another interventional clinical trial (either active or follow up phase) during the study period.
15. Participated in an A(H7) influenza vaccine study in the past or have a history of A(H7) influenza infection prior to vaccination in this study.
16. Have known human immunodeficiency virus, hepatitis B, or hepatitis C infection (based on medical history).
17. Have a history of alcohol or drug abuse in the last 5 years.
18. Have a body mass index >35 kg/m2.
19. Have a first degree relative with narcolepsy.
20. Have any laboratory test result or clinical findings (including vital signs) that singly or in combination are likely to unfavorably alter the risk-benefit of participation or to confound study safety or immunogenicity results. participants cannot be rescreened based on abnormal laboratory test results.
21. Alanine aminotransferase (AST) >2 times the upper limit of normal (ULN), or bilirubin >1.5 times the ULN unless isolated Gilbert's syndrome. participants cannot be rescreened based on abnormal laboratory test results.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 366 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Adams, MD, Principal Investigator — Central Kentucky Research; Matthew Davis, MD, Principal Investigator — Rochester Clinical Research; Carlos Fierro, MD, Principal Investigator — Johnson County Clin-Trials; Terry Poling, MD, Principal Investigator — Heartland Research Associates
Locations (4):
- United States (4):
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Rochester Clinical Research, Inc, Rochester, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 3.75 µg Panblok H7 Plus AS03: Participants dosed intramuscularly (IM) on Days 1 and 29 with 3.75 µg Panblok H7 plus AS03
- 7.5 µg Panblok H7 Plus AS03: Participants dosed intramuscularly (IM) on Days 1 and 29 with 7.5 µg Panblok H7 plus AS03
- 15 µg Panblok H7 Plus AS03: Participants dosed intramuscularly (IM) on Days 1 and 29 with 15 µg Panblok H7 plus AS03
- 3.75 µg Panblok H7 Plus MF59: Participants dosed intramuscularly (IM) on Days 1 and 29 with 3.75 µg Panblok H7 plus MF59
- 7.5 µg Panblok H7 Plus MF59: Participants dosed intramuscularly (IM) on Days 1 and 29 with 7.5 µg Panblok H7 plus MF59
- 15 µg Panblok H7 Plus MF59: Participants dosed intramuscularly (IM) on Days 1 and 29 with 15 µg Panblok H7 plus MF59
Period: Overall Study
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03 | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Started | 62 | 60 | 62 | 61 | 60 | 61
Completed | 55 | 54 | 55 | 54 | 56 | 57
Not Completed | 7 | 6 | 7 | 7 | 4 | 4
Not completed — Lost to Follow-up | 5 | 4 | 5 | 5 | 4 | 3
Not completed — Withdrawal by Subject | 2 | 2 | 2 | 1 | 0 | 1
Not completed — BARDA regulatory agency or IRB decision | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03 | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59 | Total
Number analyzed (Participants) | 62 | 60 | 62 | 61 | 60 | 61 | 366
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 2 | 1 | 0 | 0 | 3
  Between 18 and 65 years | 62 | 60 | 60 | 60 | 60 | 61 | 363
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (7.92) | 34.3 (9.14) | 35.8 (9.29) | 35 (9.58) | 37.1 (7.66) | 35.8 (8.53) | 35.4 (8.65)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 32 | 31 | 30 | 37 | 37 | 35 | 202
  Male | 30 | 29 | 32 | 24 | 23 | 26 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 7 | 1 | 2 | 4 | 22
  Not Hispanic or Latino | 60 | 54 | 55 | 60 | 58 | 57 | 344
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 0 | 2 | 0 | 4
  Asian | 1 | 1 | 0 | 0 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 17 | 8 | 9 | 13 | 5 | 60
  White | 50 | 42 | 52 | 51 | 43 | 53 | 291
  More than one race | 3 | 0 | 0 | 1 | 1 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 62 | 60 | 62 | 61 | 60 | 61 | 366

OUTCOME MEASURES:

1. Primary Outcome: Solicited Local Reactogenicity Symptoms for Participants Given Adjuvant AS03
Description: Count of participants who experienced at least one of the following during at least one of the time frames specified:
  Solicited local reactions at the injection site: erythema/redness, induration/swelling, and pain
Time Frame: Day 1-8, Day 29-36 (within 8 days of each vaccination, inclusive of the vaccination day)
Population: Safety population includes all participants who received any amount of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 62 | 60 | 62
Participants | 42 | 44 | 36

2. Primary Outcome: Solicited Systemic Reactogenicity Symptoms for Participants Given Adjuvant AS03
Description: Count of participants who experienced at least one of the following during at least one of the time frames specified:
  Solicited systemic reactions include fever, myalgia (muscle pain), arthralgia (joint pain), fatigue, headache, nausea, vomiting, diarrhea, and chills.
Time Frame: Day 1-8, Day 29-36 (within 8 days of each vaccination, inclusive of the vaccination day)
Population: Safety population includes all participants who received any amount of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 62 | 60 | 62
Participants | 25 | 28 | 27

3. Primary Outcome: Solicited Local Reactogenicity Symptoms for Participants Given Adjuvant MF59
Description: as for outcome 1
Time Frame: Day 1-8, Day 29-36 (within 8 days of each vaccination, inclusive of the vaccination day)
Population: Safety population includes all participants who received any amount of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 61 | 60 | 61
Participants | 37 | 30 | 29

4. Primary Outcome: Solicited Systemic Reactogenicity Symptoms for Participants Given Adjuvant MF59
Description: as for outcome 2
Time Frame: Day 1-8, Day 29-36 (within 8 days of each vaccination, inclusive of the vaccination day)
Population: Safety population includes all participants who received any amount of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 61 | 60 | 61
Participants | 27 | 24 | 28

5. Primary Outcome: Seroprotection Based on Serum Hemagglutination-inhibition (HAI) Antibody Titers Against Guangdong Strain for Participants Given Adjuvant AS03
Description: The percentage of participants achieving seroprotection, defined as a serum HAI antibody titer >= 1:40 against the H7 antigen (protein) contained in the vaccine. A higher HAI titer means a better immune response to the vaccine. A titer of 1:40 or greater is considered to be a sufficient amount of antibody to avoid influenza infection in half of exposed individuals.
Time Frame: Day 50
Population: Immunogenicity Per Protocol Population (IPPP) includes all participants who received a full dose of vaccine at Days 1 and 29 as assigned by randomization within protocol visit windows, had determinate assay results at Day 50 within protocol visit window, and had no major protocol deviations that may have an impact on immunogenicity assessments
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 56 | 54 | 56
Participants | 53 | 53 | 56

6. Primary Outcome: Seroprotection Based on Serum Hemagglutination-inhibition (HAI) Antibody Titers Against Guangdong Strain for Participants Given Adjuvant MF59
Description: as for outcome 5
Time Frame: Day 50
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 58 | 57 | 58
Participants | 47 | 47 | 48

7. Primary Outcome: Seroprotection Based on Serum Hemagglutination-inhibition (HAI) Antibody Titers Against the Hong Kong Strain for Participants Given Adjuvant AS03
Description: as for outcome 5
Time Frame: Day 50
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 56 | 54 | 56
Participants | 48 | 52 | 55

8. Primary Outcome: Seroprotection Based on Serum Hemagglutination-inhibition (HAI) Antibody Titers Against the Hong Kong Strain for Participants Given Adjuvant MF59
Description: as for outcome 5
Time Frame: Day 50
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 58 | 57 | 58
Participants | 37 | 35 | 47

9. Secondary Outcome: Treatment-emergent Serious Adverse Events (SAEs) for Participants Given Adjuvant AS03
Description: Count of participants who experienced at least one serious adverse event
Time Frame: Day 1 through Day 394
Population: Safety population includes all participants who received any amount of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 62 | 60 | 62
Participants | 3 | 1 | 3

10. Secondary Outcome: Treatment-emergent Serious Adverse Events (SAEs) for Participants Given Adjuvant MF59
Description: Count of participants who experienced at least one serious adverse event
Time Frame: Day 1 through Day 394
Population: Safety population includes all participants who received any amount of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 61 | 60 | 61
Participants | 1 | 2 | 0

11. Secondary Outcome: Treatment-emergent Medically Attended Adverse Events (MAAEs) for Participants Given Adjuvant AS03
Description: Count of participants who experienced at least one adverse event that requires a visit to medical personnel, including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason occurring post-vaccination.
Time Frame: Day 1 through Day 394
Population: Safety population includes all participants who received any amount of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 62 | 60 | 62
Participants | 11 | 8 | 13

12. Secondary Outcome: Treatment-emergent Medically Attended Adverse Events (MAAEs) for Participants Given Adjuvant MF59
Description: as for outcome 11
Time Frame: Day 1 through Day 394
Population: Safety population includes all participants who received any amount of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 61 | 60 | 61
Participants | 9 | 16 | 10

13. Secondary Outcome: Treatment-emergent Potentially Immune Mediated Medical Conditions (PIMMCs) for Participants Given Adjuvant AS03
Description: Count of participants who experienced at least one medical condition that was potentially immune mediated occurring post-vaccination
Time Frame: Day 1 through Day 394
Population: Safety population includes all participants who received any amount of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 62 | 60 | 62
Participants | 0 | 0 | 0

14. Secondary Outcome: Treatment-emergent Potentially Immune Mediated Medical Conditions (PIMMCs) for Participants Given Adjuvant MF59
Description: as for outcome 13
Time Frame: Day 1 through Day 394
Population: Safety population includes all participants who received any amount of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 61 | 60 | 61
Participants | 0 | 0 | 0

15. Secondary Outcome: Treatment-emergent Unsolicited Adverse Events for Participants Given Adjuvant AS03
Description: Count of participants who experienced at least one unsolicited adverse event (i.e. adverse events not included in the solicited local and systemic adverse event list nor considered a serious AE, MAAE or PIMMC ) that occur post-vaccination.
Time Frame: Day 1 through Day 53, which is the upper window of the Day 50 visit
Population: Safety population includes all participants who received any amount of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 62 | 60 | 62
Participants | 24 | 25 | 22

16. Secondary Outcome: Treatment-emergent Unsolicited Adverse Events for Participants Given Adjuvant MF59
Description: Count of participants who experienced at least one unsolicited adverse event (i.e. adverse events not included in the solicited local and systemic adverse event list nor considered a serious AE, MAAE or PIMMC) that occur post-vaccination.
Time Frame: Day 1 through Day 50
Population: Safety population includes all participants who received any amount of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 61 | 60 | 61
Participants | 24 | 24 | 21

17. Secondary Outcome: Seroprotection Based on Serum Hemagglutination-inhibition (HAI) Antibody Titers Against Guangdong Strain for Participants Given Adjuvant AS03
Description: as for outcome 5
Time Frame: Day 50
Population: The immunogenicity full analysis population (IFAP) includes all participants who were randomized, received at least one vaccination, and had determinate assay results at any post-vaccination visit. Only participants with non-missing Day 50 results are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 59 | 57 | 58
Participants | 55 | 55 | 58

18. Secondary Outcome: Seroprotection Based on Serum Hemagglutination-inhibition (HAI) Antibody Titers Against the Hong Kong Strain for Participants Given Adjuvant MF59
Description: as for outcome 5
Time Frame: Day 50
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 59 | 59 | 59
Participants | 38 | 36 | 47

19. Secondary Outcome: Seroprotection Based on Serum Hemagglutination-inhibition (HAI) Antibody Titers Against the Hong Kong Strain for Participants Given Adjuvant AS03
Description: as for outcome 5
Time Frame: Day 50
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 59 | 57 | 58
Participants | 50 | 54 | 57

20. Secondary Outcome: Serum Hemagglutination-inhibition (HAI) Antibody Titers Against the Guangdong Strain for Participants Given Adjuvant AS03
Description: Serum HAI antibody titers against the H7 antigen (protein) contained in the vaccine. A higher HAI titer means a better immune response to the vaccine.
Time Frame: Screening and Days 29, 50, 121 and 212
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 56 | 54 | 56
Titers
  Screening | 5.1 [5.0 to 5.2] | 5.3 [5.0 to 5.7] | 5.5 [5.1 to 5.9]
  Visit 4/Day 29 | 8.7 [7 to 10.8] | 12.3 [9.4 to 16] | 12.4 [9.2 to 16.8]
  Visit 7/Day 50 | 297.1 [216.5 to 407.7] | 438.3 [329.4 to 583] | 505.9 [399.7 to 640.2]
  Visit 8/Day 121 | 58.8 [43.9 to 78.8] | 73 [55.5 to 96] | 90 [70.2 to 115.3]
  Visit 9/Day 212 | 21.2 [15.6 to 28.8] | 21.6 [16.2 to 28.7] | 26 [18.9 to 35.7]

21. Secondary Outcome: Seroprotection Based on Serum Hemagglutination-inhibition (HAI) Antibody Titers Against Guangdong Strain for Participants Given Adjuvant MF59
Description: as for outcome 5
Time Frame: Day 50
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 59 | 59 | 59
Participants | 48 | 48 | 48

22. Secondary Outcome: Seroconversion Based on Serum Microneutralization (MN) Antibody Titers Against Guangdong Strain for Participants Given Adjuvant AS03
Description: The percentage of participants obtaining seroconversion based on MN antibody titers, defined as either a prevaccination MN titer <1:10 and a postvaccination MN titer ≥1:40, or a prevaccination MN titer ≥1:10 and a minimum 4 fold rise in postvaccination MN titer. Seroconversion represents the minimum intended effect of vaccination.
Time Frame: Days 29, 50, 121, and 212
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 56 | 54 | 56
Participants
  Visit 4/Day 29 | 0 | 0 | 1
  Visit 7/Day 50 | 51 | 50 | 54
  Visit 8/Day 121 | 34 | 40 | 44
  Visit 9/Day 212 | 22 | 25 | 28

23. Secondary Outcome: Serum Hemagglutination-inhibition (HAI) Antibody Titers Against the Guangdong Strain for Participants Given Adjuvant MF59
Description: as for outcome 20
Time Frame: Screening and Days 29, 50, 121 and 212
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 58 | 57 | 58
Titers
  Screening | 5.1 [5 to 5.2] | 5.5 [5 to 6.1] | 5.1 [5 to 5.2]
  Visit 4/Day 29 | 6.1 [5.1 to 7.3] | 6.6 [5.7 to 7.7] | 6.4 [5.6 to 7.3]
  Visit 7/Day 50 | 76.3 [55.9 to 104] | 106.5 [74.1 to 153] | 130.6 [93.1 to 183.2]
  Visit 8/Day 121 | 18.1 [13.6 to 24.1] | 20.7 [14.9 to 28.8] | 33.2 [25.1 to 43.9]
  Visit 9/Day 212 | 6.8 [6 to 7.7] | 8.9 [7.1 to 11.1] | 11.4 [8.7 to 15]

24. Secondary Outcome: Serum Hemagglutination-inhibition (HAI) Antibody Titers Against the Guangdong Strain for Participants Given Adjuvant MF59
Description: as for outcome 20
Time Frame: Day 50
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 59 | 59 | 59
Titers | 75.4 [55.6 to 102.4] | 103 [72.1 to 147.2] | 124.3 [87.9 to 175.8]

25. Secondary Outcome: Serum Hemagglutination-inhibition (HAI) Antibody Titers Against the Hong Kong Strain for Participants Given Adjuvant AS03
Description: as for outcome 20
Time Frame: Screening and Days 29, 50, 121 and 212
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 56 | 54 | 56
Titers
  Screening | 5 [5 to 5] | 5.2 [4.9 to 5.6] | 5.2 [5 to 5.4]
  Visit 4/Day 29 | 5.9 [5.2 to 6.7] | 8.3 [6.7 to 10.3] | 8.4 [6.6 to 10.7]
  Visit 7/Day 50 | 170.2 [119.9 to 241.7] | 302 [218.9 to 416.7] | 316.7 [246.2 to 407.4]
  Visit 8/Day 121 | 45.2 [33.4 to 61.1] | 57.7 [42.5 to 78.4] | 69.7 [53.1 to 91.6]
  Visit 9/Day 212 | 25 [18.3 to 34.2] | 28.1 [20.1 to 39.2] | 32.9 [24.4 to 44.4]

26. Secondary Outcome: Serum Hemagglutination-inhibition (HAI) Antibody Titers Against the Hong Kong Strain for Participants Given Adjuvant AS03
Description: as for outcome 20
Time Frame: Day 50
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 59 | 57 | 58
Titers | 163.8 [115.7 to 231.9] | 274.9 [195.3 to 386.9] | 313.1 [243.1 to 403.1]

27. Secondary Outcome: Serum Hemagglutination-inhibition (HAI) Antibody Titers Against the Hong Kong Strain for Participants Given Adjuvant MF59
Description: as for outcome 20
Time Frame: Screening and Days 29, 50, 121 and 212
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 58 | 57 | 58
Titers
  Screening | 5.1 [5 to 5.2] | 5.1 [5 to 5.2] | 5.3 [4.8 to 5.8]
  Visit 4/Day 29 | 5.7 [5.1 to 6.3] | 5.6 [5.1 to 6.1] | 5.6 [5.2 to 6.1]
  Visit 7/Day 50 | 47.6 [33.7 to 67.1] | 60.5 [40.5 to 90.4] | 74.5 [53.3 to 104]
  Visit 8/Day 121 | 13 [10.2 to 16.6] | 15.1 [11.2 to 20.4] | 20.9 [15.6 to 27.8]
  Visit 9/Day 212 | 7.8 [6.7 to 9.1] | 11.3 [8.6 to 14.8] | 13.6 [10.1 to 18.2]

28. Secondary Outcome: Serum Hemagglutination-inhibition (HAI) Antibody Titers Against the Hong Kong Strain for Participants Given Adjuvant MF59
Description: as for outcome 20
Time Frame: Day 50
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 59 | 59 | 59
Titers | 47.4 [33.8 to 66.5] | 58.6 [39.4 to 87.2] | 71.1 [50.6 to 100]

29. Secondary Outcome: Seroprotection Based on Serum Hemagglutination-inhibition (HAI) Antibody Titers Against Guangdong Strain for Participants Given Adjuvant AS03
Description: as for outcome 5
Time Frame: Screening, Day 29, Day 121, Day 212
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 56 | 54 | 56
Participants
  Screening | 0 | 0 | 0
  Visit 4/Day 29 | 7 | 10 | 13
  Visit 8/Day 121 | 40 | 45 | 47
  Visit 9/Day 212 | 21 | 19 | 23

30. Secondary Outcome: Seroprotection Based on Serum Hemagglutination-inhibition (HAI) Antibody Titers Against Guangdong Strain for Participants Given Adjuvant MF59
Description: as for outcome 5
Time Frame: Screening, Day 29, Day 121, Day 212
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 58 | 57 | 58
Participants
  Screening | 0 | 0 | 0
  Visit 4/Day 29 | 1 | 3 | 0
  Visit 8/Day 121 | 19 | 24 | 34
  Visit 9/Day 212 | 1 | 4 | 7

31. Secondary Outcome: Seroprotection Based on Serum Hemagglutination-inhibition (HAI) Antibody Titers Against Hong Kong Strain for Participants Given Adjuvant AS03
Description: as for outcome 5
Time Frame: Screening, Day 29, Day 121, Day 212
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 56 | 54 | 56
Participants
  Screening | 0 | 0 | 0
  Visit 4/Day 29 | 2 | 5 | 4
  Visit 8/Day 121 | 37 | 40 | 45
  Visit 9/Day 212 | 22 | 22 | 26

32. Secondary Outcome: Seroprotection Based on Serum Hemagglutination-inhibition (HAI) Antibody Titers Against Hong Kong Strain for Participants Given Adjuvant MF59
Description: as for outcome 5
Time Frame: Screening, Day 29, Day 121, Day 212
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 58 | 57 | 58
Participants
  Screening | 0 | 0 | 1
  Visit 4/Day 29 | 1 | 0 | 0
  Visit 8/Day 121 | 10 | 15 | 22
  Visit 9/Day 212 | 1 | 8 | 11

33. Secondary Outcome: Seroconversion Based on Serum Hemagglutination-inhibition (HAI) Antibody Titers Against Guangdong Strain for Participants Given Adjuvant AS03
Description: The percentage of participants obtaining seroconversion based on HAI antibody titers, defined as either a prevaccination HAI titer <1:10 and a postvaccination HAI titer ≥1:40, or a prevaccination HAI titer ≥1:10 and a minimum 4 fold rise in postvaccination HAI titer. Seroconversion represents the minimum intended effect of vaccination.
Time Frame: Day 29, Day 50, Day 121, Day 212
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 56 | 54 | 56
Participants
  Visit 4/Day 29 | 7 | 10 | 12
  Visit 7/Day 50 | 53 | 53 | 56
  Visit 8/Day 121 | 40 | 45 | 47
  Visit 9/Day 212 | 21 | 19 | 23

34. Secondary Outcome: Seroconversion Based on Serum Hemagglutination-inhibition (HAI) Antibody Titers Against Guangdong Strain for Participants Given Adjuvant MF59
Description: as for outcome 33
Time Frame: Day 29, Day 50, Day 121, Day 212
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 58 | 57 | 58
Participants
  Visit 4/Day 29 | 1 | 2 | 0
  Visit 7/Day 50 | 47 | 47 | 48
  Visit 8/Day 121 | 19 | 23 | 34
  Visit 9/Day 212 | 1 | 4 | 7

35. Secondary Outcome: Seroconversion Based on Serum Hemagglutination-inhibition (HAI) Antibody Titers Against Hong Kong Strain for Participants Given Adjuvant AS03
Description: as for outcome 33
Time Frame: Day 29, Day 50, Day 121, Day 212
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 56 | 54 | 56
Participants
  Visit 4/Day 29 | 2 | 5 | 4
  Visit 7/Day 50 | 48 | 52 | 55
  Visit 8/Day 121 | 37 | 39 | 45
  Visit 9/Day 212 | 22 | 22 | 26

36. Secondary Outcome: Seroconversion Based on Serum Hemagglutination-inhibition (HAI) Antibody Titers Against Hong Kong Strain for Participants Given Adjuvant MF59
Description: as for outcome 33
Time Frame: Day 29, Day 50, Day 121, Day 212
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 58 | 57 | 58
Participants
  Visit 4/Day 29 | 1 | 0 | 0
  Visit 7/Day 50 | 37 | 35 | 47
  Visit 8/Day 121 | 10 | 15 | 21
  Visit 9/Day 212 | 1 | 8 | 11

37. Secondary Outcome: Seroconversion Based on Serum Microneutralization (MN) Antibody Titers Against Guangdong Strain for Participants Given Adjuvant MF59
Description: as for outcome 22
Time Frame: Day 29, Day 50, Day 121, Day 212
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 58 | 57 | 58
Participants
  Visit 4/Day 29 | 0 | 0 | 0
  Visit 7/Day 50 | 40 | 39 | 44
  Visit 8/Day 121 | 11 | 14 | 21
  Visit 9/Day 212 | 2 | 4 | 11

38. Secondary Outcome: Seroconversion Based on Serum Microneutralization (MN) Antibody Titers Against Hong Kong Strain for Participants Given Adjuvant AS03
Description: as for outcome 22
Time Frame: Day 29, Day 50, Day 121, Day 212
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 56 | 54 | 56
Participants
  Visit 4/Day 29 | 0 | 2 | 7
  Visit 7/Day 50 | 53 | 53 | 56
  Visit 8/Day 121 | 38 | 43 | 47
  Visit 9/Day 212 | 25 | 28 | 34

39. Secondary Outcome: Seroconversion Based on Serum Microneutralization (MN) Antibody Titers Against Hong Kong Strain for Participants Given Adjuvant MF59
Description: as for outcome 22
Time Frame: Day 29, Day 50, Day 121, Day 212
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 58 | 57 | 58
Participants
  Visit 4/Day 29 | 1 | 1 | 0
  Visit 7/Day 50 | 46 | 44 | 47
  Visit 8/Day 121 | 11 | 21 | 27
  Visit 9/Day 212 | 3 | 6 | 15

40. Secondary Outcome: Serum Hemagglutination-inhibition (HAI) Antibody Titers Against the Guangdong Strain for Participants Given Adjuvant AS03
Description: as for outcome 20
Time Frame: Day 50
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 59 | 57 | 58
Titers | 276.3 [200.1 to 381.5] | 400.7 [291.9 to 550.1] | 489.1 [383 to 624.5]

41. Secondary Outcome: Serum Microneutralization (MN) Antibody Titers Against the Guangdong Strain for Participants Given Adjuvant AS03
Description: Serum MN antibody titers against the H7 antigen (protein) contained in the vaccine. A higher MN titer means a better immune response to the vaccine.
Time Frame: Screening and Days 29, 50, 121 and 212
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 56 | 54 | 56
Titers
  Screening | 5.0 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  Visit 4/Day 29 | 5.3 [5 to 5.5] | 6.2 [5.6 to 6.9] | 6.3 [5.5 to 7.2]
  Visit 7/Day 50 | 201.2 [147.4 to 274.6] | 274.3 [197.4 to 381.2] | 286.3 [218.1 to 375.7]
  Visit 8/Day 121 | 51.4 [40.8 to 64.7] | 58.1 [44.6 to 75.6] | 66.6 [53.4 to 83.1]
  Visit 9/Day 212 | 29 [22.2 to 38] | 29.7 [22.7 to 38.8] | 34.4 [27.6 to 42.9]

42. Secondary Outcome: Serum Microneutralization (MN) Antibody Titers Against the Guangdong Strain for Participants Given Adjuvant MF59
Description: as for outcome 20
Time Frame: Screening and Days 29, 50, 121 and 212
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 58 | 57 | 58
Titers
  Screening | 5.1 [5 to 5.1] | 5 [5 to 5.1] | 5 [5 to 5]
  Visit 4/Day 29 | 5.2 [4.9 to 5.5] | 5 [5 to 5.1] | 5.2 [4.9 to 5.4]
  Visit 7/Day 50 | 53 [39.9 to 70.3] | 67.1 [46.3 to 97.1] | 81.9 [60.1 to 111.7]
  Visit 8/Day 121 | 15.1 [12.2 to 18.8] | 18.5 [14.5 to 23.5] | 25.6 [19.7 to 33.1]
  Visit 9/Day 212 | 8.2 [7 to 9.7] | 10.7 [8.9 to 13] | 14 [10.8 to 18]

43. Secondary Outcome: Serum Microneutralization (MN) Antibody Titers Against the Hong Kong Strain for Participants Given Adjuvant AS03
Description: as for outcome 20
Time Frame: Screening and Days 29, 50, 121 and 212
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3.75 µg Panblok H7 Plus AS03 | 7.5 µg Panblok H7 Plus AS03 | 15 µg Panblok H7 Plus AS03
Number analyzed (Participants) | 56 | 54 | 56
Titers
  Screening | 5 [5 to 5.1] | 5 [5 to 5] | 5.2 [4.9 to 5.4]
  Visit 4/Day 29 | 6.4 [5.7 to 7.3] | 7.8 [6.7 to 9.1] | 8.9 [7.2 to 11.2]
  Visit 7/Day 50 | 256.1 [190.3 to 344.6] | 326.2 [238.1 to 446.9] | 394.9 [303.8 to 513.4]
  Visit 8/Day 121 | 58.4 [44.9 to 76] | 71.6 [53.6 to 95.6] | 95.4 [73.3 to 124.4]
  Visit 9/Day 212 | 31.5 [23.7 to 41.9] | 34.4 [26.1 to 45.4] | 41.1 [32 to 52.7]

44. Secondary Outcome: Serum Microneutralization (MN) Antibody Titers Against the Hong Kong Strain for Participants Given Adjuvant MF59
Description: as for outcome 20
Time Frame: Screening and Days 29, 50, 121 and 212
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 3.75 µg Panblok H7 Plus MF59 | 7.5 µg Panblok H7 Plus MF59 | 15 µg Panblok H7 Plus MF59
Number analyzed (Participants) | 58 | 57 | 58
Titers
  Screening | 5.1 [5 to 5.2] | 5.3 [5 to 5.6] | 5.1 [5 to 5.1]
  Visit 4/Day 29 | 5.8 [5.2 to 6.5] | 6 [5.3 to 6.7] | 5.9 [5.4 to 6.4]
  Visit 7/Day 50 | 67.3 [51.4 to 88] | 87.1 [59.8 to 126.9] | 113.8 [80.4 to 161.1]
  Visit 8/Day 121 | 15.7 [12.5 to 19.8] | 20 [15 to 26.6] | 27.1 [20 to 36.7]
  Visit 9/Day 212 | 8.7 [7.3 to 10.5] | 11.5 [9.2 to 14.4] | 15.2 [11.6 to 19.9]

ADVERSE EVENTS:
Time Frame: 13 months
Arm/Group | 3.75 ug Panblok H7 Plus AS03 | 7.5 ug Panblok H7 Plus AS03 | 15 ug Panblok H7 Plus AS03 | 3.75 ug Panblok H7 Plus MF59 | 7.5 ug Panblok H7 Plus MF59 | 15 ug Panblok H7 Plus MF59
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/60 | 0/62 | 0/61 | 0/60 | 0/61
Serious Adverse Events (participants affected / at risk) | 3/62 | 1/60 | 3/62 | 1/61 | 2/60 | 0/61
Other Adverse Events (participants affected / at risk) | 48/62 | 47/60 | 40/62 | 47/61 | 40/60 | 42/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3.75 ug Panblok H7 Plus AS03 (N=62) | 7.5 ug Panblok H7 Plus AS03 (N=60) | 15 ug Panblok H7 Plus AS03 (N=62) | 3.75 ug Panblok H7 Plus MF59 (N=61) | 7.5 ug Panblok H7 Plus MF59 (N=60) | 15 ug Panblok H7 Plus MF59 (N=61)
Cardiac septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary artery stenosis congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colloid brain cyst (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Monoplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3.75 ug Panblok H7 Plus AS03 (N=62) | 7.5 ug Panblok H7 Plus AS03 (N=60) | 15 ug Panblok H7 Plus AS03 (N=62) | 3.75 ug Panblok H7 Plus MF59 (N=61) | 7.5 ug Panblok H7 Plus MF59 (N=60) | 15 ug Panblok H7 Plus MF59 (N=61)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 5 (7) | 9 (12) | 9 (10) | 10 (15) | 8 (9)
Nausea (Gastrointestinal disorders) | 7 (9) | 7 (11) | 10 (10) | 12 (18) | 4 (5) | 9 (9)
Chills (General disorders) | 7 (8) | 7 (10) | 6 (6) | 6 (7) | 5 (5) | 4 (4)
Fatigue (General disorders) | 17 (22) | 15 (18) | 19 (24) | 16 (22) | 11 (13) | 10 (11)
Injection site erythema (General disorders) | 5 (5) | 7 (8) | 3 (4) | 7 (8) | 2 (2) | 2 (2)
Injection site induration (General disorders) | 3 (4) | 8 (11) | 6 (9) | 7 (9) | 2 (2) | 1 (1)
Injection site pain (General disorders) | 42 (70) | 42 (68) | 36 (60) | 32 (44) | 29 (42) | 29 (45)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 4 (4) | 2 (3) | 6 (7) | 6 (6) | 4 (5)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 4 (5) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 6 (8) | 6 (6) | 8 (10) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (20) | 19 (27) | 18 (24) | 16 (23) | 8 (10) | 13 (17)
Headache (Nervous system disorders) | 21 (29) | 17 (26) | 16 (23) | 16 (20) | 16 (28) | 15 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 2 (2) | 4 (5) | 3 (3) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT03283319/Prot_002.pdf
  • Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/19/NCT03283319/SAP_003.pdf